CLINICAL TRIAL: NCT04861727
Title: Use of Technology to Optimize Hypertension Treatment in Elderly People in Primary Care
Acronym: MINOR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Bahia (Other)
Responsible Party: Principal Investigator, Márcio Galvão Guimarães de Oliveira, Clinical Professor of Pharmacy and Evidence-based Health Care, Federal University of Bahia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: FARMRPA 01.2021
Record Dates: First submitted 2021-04-13; First posted 2021-04-27 (Actual); Last update posted 2022-10-05 (Actual); Status verified 2022-10

CONDITIONS: Systemic Arterial Hypertension; Pharmacotherapy; Pharmaceutical Care
Keywords: Systemic Arterial Hypertension;; Technology Applied to Health Care;; Pharmacotherapy;; Pharmaceutical Care.
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: The Control Group will be attended by Pharmacists and will have the data collected according to the standard collection instrument, will receive general guidance on blood pressure control and pharmacotherapy assessment. The Intervention Group, in addition to the control group procedures, will also perform the MRPA, the result of which will guide the pharmaceutical suggestions, when necessary, they also received a Letter of Referral to the Prescriber containing pharmaceutical suggestions for optimization of pharmacotherapy, considering the current clinical protocols.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group control (No Intervention): will be attended by Pharmacists and will have the data collected according to the standard collection instrument, will make MRPA and will receive the report and general guidance on blood pressure control and pharmacotherapy assessment
- Intervention group (Active Comparator): will be attended by Pharmacists and will have the data collected according to the standard collection instrument, will receive general guidance on blood pressure control and pharmacotherapy assessment, will also do MRPA whose result will guide pharmaceutical suggestions, when necessary, they will also receive a Referral Letter to the Prescriber containing pharmaceutical suggestions for optimization of pharmacotherapy, considering the current clinical protocols.
  Interventions: Other: MRPA procedure; Other: Pharmaceutical intervention

INTERVENTIONS:
Other: MRPA procedure — The patient will receive the device for BP measurement at home for a week and two daily measurements will be taken, one in the morning (between 6 and 10 am) and one in the afternoon / evening (between 6 pm and 10 pm), for seven days. At the end of the procedure, it is expected to record 14 measurements (representing a total of 42 in seven days), but it is considered feasible when at least 10 results are recorded, respecting the number of two measurements per day, in the periods oriented. Participants who do not reach the satisfactory number of measures or do not check between the times mentioned above, will be invited to repeat the procedure
  Arms: Intervention group
Other: Pharmaceutical intervention — The suggestion procedure, for this research, is defined as the pharmaceutical act of forwarding a letter of suggestion to the prescriber, previously agreed with the patient, based on clinical evaluation, review of pharmacotherapy, adherence to treatment and result of the MRPA procedure.
  Arms: Intervention group

SUMMARY:
The control of blood pressure (BP) in the elderly is influenced by several factors, among them, the measurement methodology. The measurement of BP in the office is prone to failures, so the use of technology associated with blood pressure measurements at home is an alternative to minimize failures and contribute to the optimization of treatment. The objective of this study will be to evaluate the adequacy of the treatment of Systemic Arterial Hypertension (SAH) in primary care using Home Blood Pressure Monitoring (MRPA). Method: Randomized clinical trial with hypertensive patients, aged 60 years or over, attended at the Family Pharmacy service inserted in the primary care of the municipal health network. The subjects who accept to participate in the study will be randomized to the intervention / control groups. submitted to MRPA, will undergo analysis of the pharmacotherapy prescribed for the treatment of SAH, collection of clinical data, which together will support the assessment of the adequacy of the treatment of hypertension. When inadequacies in pharmacotherapy are identified, suggestions for changes will be forwarded to the prescriber / professional or assistant health team, weighted by the pharmacist in agreement with the patient and according to the guidelines of the Brazilian Guideline on Hypertension. The outcomes: changes in treatment and blood pressure control in the intervention and control groups will be evaluated.

DETAILED DESCRIPTION:
The study will be carried out at a municipal public pharmacy. The subjects will be users of the Family Pharmacy, aged 60 years or over, who seek the service to remove the drugs prescribed for the treatment of Systemic Arterial Hypertension. In order to calculate the sample for this study, the incidence of patients with Hypertension System who need treatment adjustments (under- or over-treatment) will be considered. It is expected that in the intervention group, MRPA indicates that 30% of patients will need to change their pharmacotherapy and, in the control group, using the office measure, 10%. For a two-tailed test with 80% power, 5% sampling error and 95% confidence level, the sample will be 160 users in the intervention group and 160 in the control group. Considering the pandemic of COVID-19 and the risk of infection during care in health services, whether from patients or health professionals from the health care network, the Family Pharmacy already adopts the screening for respiratory symptoms that identify suspected infection by Sars-Cov-2.To minimize the impact of selection and information bias, the following procedure will be used to select individuals: during attendance at the windows, each trained attendant will invite patients with eligibility criteria, when they accept, they will be inserted in the service schedule. The selection for control group and intervention group will take place by drawing from the list of scheduled people, with 3 participants being drawn for the Intervention Group, totaling 160 participants in each group. Data collection will only occur after signing the Informed Consent Form (ICF). The Control Group will be attended by Pharmacists and will have the data collected according to the standard collection instrument, will receive general guidance on blood pressure control and pharmacotherapy assessment. The Intervention Group, in addition to the control group procedures, will also perform the MRPA, the result of which will guide the pharmaceutical suggestions, when necessary, they also received a Letter of Referral to the Prescriber containing pharmaceutical suggestions for optimization of pharmacotherapy, considering the current clinical protocols. In the service, patients and companions will be instructed on preventive measures against Sars-coV-2 infection, in addition to performing hand hygiene with water and liquid soap or 70% alcohol gel. The office will undergo cleaning before and after use, as well as the material, in addition to adopting the time of 15 minutes between appointments, maintaining the ventilation of the room, following all the recommendations of the Ministry of Health. Pharmaceutical evaluation is already a routine of the service. For the purposes of this research, the procedures will be added to standardized instruments and routines to guarantee methodological quality and answer the questions of this research. The Data Collection Form (Appendix I) will be used, which includes the collection of data related to sociodemographic and clinical characteristics. In order to assess adherence, the Portuguese version of the Brief Medication Questionnaire (BMQ) will be used in two stages: during the initial evaluation, when the patient was included in the research and 45 days after the intervention.

The pharmaceutical suggestion procedure, for this research, is defined as forwarding a letter of suggestion to the prescriber, previously agreed with the patient, based on clinical evaluation, review of pharmacotherapy, adherence to treatment and result of the MRPA procedure. The definition of the conducts to be adopted will be based on the 8th Brazilian Guideline on Systemic Arterial Hypertension, and in a complementary way - as it is an elderly patient (60 years old or more) - by the Brazilian Consensus on Potential Medicines Inappropriate for the Elderly.

The data will be tabulated and analyzed using the SPPS® Statistic 25 software. The Kolmogorov-Sminorv test will be used to assess the data distribution. The paired T test will be used to assess the differences between BP measurements in the office and the MRPA mean. Continuous variables with normal distribution will be presented as means, standard deviations and Odds Ratio. Categorical variables will be presented as a proportion, using the Chi-square test. Values of p <0.05 will be considered significant.

To compare the proportion of patients with controlled and uncontrolled blood pressure, before and after application of the intervention, the chi-square test (χ2) will be used. Mean or median values of the MRPA Blood Pressure Mean will also be compared before and after the intervention / description and adherence before and after the MRPA procedure (baseline and at the end of the study) using the paired T test or Wilcoxon.

ELIGIBILITY:
Inclusion Criteria:

* Elderly with confirmation of a diagnosis of arterial hypertension (self-report, based on medical report or prescription)
* Using antihypertensive pharmacotherapy

Exclusion Criteria:

* Users who, for whatever reason, are unable to perform MRPA.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2021-06-06 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Change in Mean Blood Pressure in MRPA | 45 days after the intervention
  Change from baseline systolic blood pressure in 45 days

SECONDARY OUTCOMES:
Proportion of patients identified with undertreatment | Baseline
  Patients who had blood pressure above target, needing to add doses or more antihypertensive drugs in pharmacotherapy
Proportion of patients identified with overtreatment | Baseline
  Patients who had blood pressure below the target, needing to prescribe doses or withdraw antihypertensive drugs from pharmacotherapy
Number of drug deprescribing suggestions made | Baseline
  Deprescribing suggestions made by pharmacists based on the average blood pressure value and clinical treatment protocols
Number of pharmacotherapy adequacy suggestions accepted by the prescriber | 45 days after the intervention
  Number of pharmacotherapy adequacy suggestions accepted by the prescriber

CONTACTS AND LOCATIONS:
Overall Officials: Marcio GG Oliveira, Principal Investigator — Federal University of Bahia
Locations (1):
- Farmácia Escola da UFBA, campus Anísio Teixeira, Vitória da Conquista, Estado de Bahia, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Silva IM, Moreira PM, Santos AM, Castro PR, Aguiar EC, Oliveira MG. Desprescribing antihypertensives in older people in primary care: subgroup analysis of the MINOR randomised clinical trial. Int J Clin Pharm. 2025 Feb;47(1):53-59. doi: 10.1007/s11096-024-01805-y. Epub 2024 Nov 6. PMID 39503798
- [Derived] Moreira PM, Aguiar EC, Castro PR, Almeida KC, Dourado JA, Paula SM, Melo MF, Santos PM, Oliveira MG. Optimizing Hypertension Treatment in Older Patients Through Home Blood Pressure Monitoring by Pharmacists in Primary Care: The MINOR Clinical Trial. Clin Ther. 2023 Oct;45(10):941-946. doi: 10.1016/j.clinthera.2023.06.007. Epub 2023 Jun 24. PMID 37365046